CLINICAL TRIAL: NCT00165815
Title: The Efficacy, Tolerability and Safety of Donepezil (Aricept) in Parkinson's Disease Patients With Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2020-E044-316
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2005-11

CONDITIONS: Dementia With Parkinson's Disease
MeSH Terms: interventions — Donepezil

INTERVENTIONS:
Drug: ARICEPT

SUMMARY:
A randomised, double-blind, 3-arm parallel group study comparing Aricept® with placebo.

ELIGIBILITY:
Patients with an established diagnosis of PD and dementia, who fulfill all of the inclusion criteria and none of the exclusion criteria listed below, will be eligible for enrolment into this study.

Best efforts must be made on clinical grounds to exclude patients with DLB and AD. The key inclusion criteria in this respect is the onset of dementia documented to have occurred at least 1 year after the diagnosis of PD.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2002-08; Study Completion 2005-07

PRIMARY OUTCOMES:
PD patients with dementia will be screened up to 4 weeks prior to initiating dose administration. Baseline measurement on efficacy measures will be conducted at baseline, after which the first dose of study medication will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Jina Schwartz, Study Director — Eisai Limited
Locations (4):
- Germany (2):
  - Allgemeines Krankenhaus Barmbeck, Hamburg, Hambug
  - Parkinson Klinik Wolfach, Wolfach, Wolfach
- Ireland (2):
  - Belfast City Hospital, Belfast, Belfast
  - Unit 20 Black Poo Technology Centerl, Blackpool, Blackpool